CLINICAL TRIAL: NCT00432094
Title: Autologous Peripheral Blood Stem Cell Transplant for Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006LS032; UMN-MT2005-21 (Other: Blood and Marrow Transplantation Program); UMN-0608M90586 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Childhood Germ Cell Tumor; Ovarian Cancer; Teratoma
Keywords: childhood extragonadal germ cell tumor; childhood malignant ovarian germ cell tumor; childhood malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; testicular choriocarcinoma and seminoma; testicular embryonal carcinoma and seminoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor; testicular seminoma; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; stage I extragonadal non-seminomatous germ cell tumor; stage I extragonadal seminoma; stage II extragonadal non-seminomatous germ cell tumor; stage II extragonadal seminoma; stage III extragonadal non-seminomatous germ cell tumor; stage III extragonadal seminoma; stage II ovarian germ cell tumor; stage I malignant testicular germ cell tumor; stage II malignant testicular germ cell tumor; adult teratoma; childhood teratoma; testicular immature teratoma; testicular mature teratoma; adult central nervous system germ cell tumor; childhood central nervous system germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Teratoma; Ovarian Germ Cell Cancer; Testicular Neoplasms; Seminoma; Endodermal Sinus Tumor; Carcinoma, Embryonal | interventions — Carboplatin; Etoposide; Ifosfamide; Paclitaxel; Thiotepa; Mesna; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: This trial is single arm study and it is non-randomized. Overall, if patients did not have enough cells to do two transplants then they only received one transplants.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 Transplants/1 Transplant (Overall) (Experimental): 2 Transplants: Patients with Germ Cell Tumors (GCT) treated with a second tandem autologous stem cell transplant (AuSCT) with non-cross-resistant conditioning regimens.
  1 Transplants:Patients with Germ cell tumors who receive one transplant only.
  Interventions: Drug: carboplatin; Drug: etoposide; Drug: ifosfamide; Drug: paclitaxel; Drug: thiotepa; Procedure: autologous hematopoietic stem cell transplantation; Drug: Mesna; Biological: filgrastim

INTERVENTIONS:
Drug: carboplatin — Days -6, -5, -4: 500mg/m2^/day intravenously (IV) over 60 minutes
Drug: etoposide — 600mg/m^2/day intravenously (IV) over 60 minutes on Days -6 through -3.
  Other Names: VP-16; Toposar
Drug: ifosfamide — 2500 mg/m^2/day continuous infusion intravenously on Days -6, -5 and -4.
  Other Names: Mitoxana; Ifex
Drug: paclitaxel — 225 mg/m^2 intravenous over 3 hours on Day -7.
  Other Names: Taxol
Drug: thiotepa — 150mg/m^2/day intravenously IV over 30 minutes; Days -6, -5 and -4
  Other Names: N,N'N'-triethylenethiophosphoramide
Procedure: autologous hematopoietic stem cell transplantation — Peripheral blood stem cell infusion (< 4 x 10^6 CD34+ cells/kg)
  Other Names: PBSC
Drug: Mesna — 2500 mg/m^2/day continuous infusion intravenously on Days -6, -5 and -4.
  Other Names: Uromitexan®
Biological: filgrastim — Beginning Day 5, G-CSF 5 μg/kg/day until absolute neutrophil count (ANC) ≥ 1500/UL for 3 consecutive days.
  Other Names: G-CSF

SUMMARY:
RATIONALE: Germ cell tumors (GCT) are highly sensitive to chemotherapy such that even with metastatic disease at diagnosis, many patients can be cured. Patients who fall into the poor risk category or others who relapse can be successfully salvaged with high dose chemotherapy and autologous stem cell transplant (AuSCT). As in other diseases such as myeloma, sequential high dose chemotherapy and AuSCT may improve overall and disease free survival.

PURPOSE: Because prior investigations in GCT suggest that a subset of high risk or relapsed patients may be cured with sequential cycles of high dose chemotherapy and AuSCT, we propose investigating how well non-cross resistant conditioning regimens work in treating patients with relapsed or high risk GCT.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine overall survival (OS) of patients with germ cell tumors treated with tandem autologous stem cell transplantation with non-cross-resistant conditioning regimens.

Secondary

* Determine disease-free survival (DFS) of patients treated with this regimen.
* Determine the toxicity of tandem transplants
* Determine the time to engraftment of neutrophils and platelets in patients treated for each transplant
* Determine the number of patients unable to adequately mobilize sufficient peripheral blood stem cells (PBSC) for tandem transplantation.
* Identify prognostic factors of patients unlikely to mobilize sufficient PBSC for tandem transplantation.
* Compare OS and DFS of patients undergoing single vs tandem transplantation.

OUTLINE:

* Peripheral blood stem cell (PBSC) mobilization with filgrastim (G-CSF): Patients receive G-CSF subcutaneously (SC) beginning on day 1 and continuing until stem cell collection is complete. Patients undergo stem cell collection beginning on day 5 of G-CSF administration and continuing for at least 3 collections until the collection goal is met.
* Second PBSC mobilization with chemotherapy: Patients not meeting the collection goal receive cyclophosphamide IV over 2 hours on day 1 and G-CSF SC beginning on day 4 and continuing until stem cell collection is complete. Patients meeting the collection goal after PBSC mobilization via G-CSF alone or in combination with chemotherapy will undergo tandem autologous transplantation. If collection goal is not met but the patient has collected > or = 2 x 10^6 CD34 cells/kg, a single autologous transplant will be performed.
* Single stem cell transplantation (SCT): Patients receive paclitaxel IV over 3 hours on day -7 and ifosfamide IV on days -6 to -4. Patients undergo reinfusion of stem cells on day 0. Patients also receive G-CSF SC or IV beginning on day 1 and continuing until blood counts recover.
* Tandem SCT: Patients receive treatment as in single SCT. Beginning 30-90 days later, patients receive carboplatin IV over 60 minutes and thiotepa IV over 30 minutes on days -6 to -4 and etoposide IV over 60 minutes on days -6 to -3. Patients undergo reinfusion of stem cells on day 0. Patients also receive G-CSF SC or IV beginning on day 5 and continuing until blood counts recover.

After completion of study treatment, patients are followed at 6, 9, and 12 months and then every 6 months for up to 2 years.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Poor Prognosis Non-Seminomas Germ Cell Tumor in ≥ PR1/CR1 or Good or Intermediate Prognosis Seminomas and Non- Seminomas Germ Cell Tumor in ≥ PR1 or ≥ CR2 as defined by the International Germ Cell Cancer Consensus Classification. Patients with increasing tumor markers only (i.e. no imaging evidence of progressive disease) are eligible for transplant.
* Age: ≥ 10 years and < 70 years of age.
* Performance status: Karnofsky ≥ 80% (subjects ≥ 16 years of age) Lansky ≥ 80% for subject 10 - 15 years of age
* Life expectancy: Greater than 8 weeks.
* Patients must have normal organ function as defined below:

  * Hematologic:

    * Hemoglobin > 8 gm/dL without transfusion and off erythropoietin for 14 days or Aranesp for 21 days
    * White blood cells (WBC) > 2.5 x 10^9/L with an absolute neutrophile count (ANC) > 1.5 x 10^9/L and off G-CSF or GM-CSF for 10 days or Neulasta for 21 days
    * Platelets > 100 x 10^9/L without transfusion and/or a bone marrow cellularity of ≥ 20%
  * Renal: Creatinine ≤ 2.0 mg/dl or creatinine clearance > 50 ml/min.
  * Hepatic: Total bilirubin ≤ 2.0 mg/dl, AST and alkaline phosphatase < 5 x upper limit of normal. No history of severe prior or ongoing chronic liver disease.
  * Cardiac: Patients must be free of symptoms of uncontrolled cardiac disease including unstable angina, decompensated congestive heart failure, or arrhythmia. LVEF ≥45% by MUGA/ECHO.
  * Pulmonary: Patients must have no significant obstructive airways disease (FEV1 must be ≥ 50% of predicted) and must have acceptable diffusion capacity (corrected DLCO > 50% of predicted).
* Patients with a history of CNS tumor involvement are eligible if they have completed treatment for CNS disease (radiotherapy or surgery or chemotherapy), have recovered from or stabilization of the side effects associated with the therapy and have no evidence of progressive CNS disease at the time of enrollment.

Exclusion Criteria:

* Patients with serious uncontrolled infections will not be eligible.
* Male and female patients of reproductive potential must use an approved contraceptive method if appropriate (for example, intrauterine device [IUD], birth control pills, or barrier device) during and for the duration of study participation. The drugs used in this study are pregnancy category D - clear evidence of risk in pregnancy.
* Pregnant and breast feeding women will not be eligible.

Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Additional Eligibility prior to Transplant Two:

* Total Collection of ≥ 4 x 10^6 CD34 cells/kg prior to transplant one
* Transplant able to occur between day +30 and day +90 from transplant one
* Recovery of blood counts as demonstrated by:

  * WBC > 2.5 x 10^9/L with an ANC > 1.5 x 10^9/L and off G-CSF for 3 days
  * Platelets > 50 x 10^9/L without transfusion in the prior 7 days
  * Renal: Creatinine ≤ 2.0 mg/dl or creatinine clearance > 50 ml/min
  * Hepatic: Total bilirubin ≤ 2.0 mg/dl, AST and alkaline phosphatase < 5 x upper limit of normal
* Infection: Patients with serious uncontrolled infections at the time of planned transplant will be excluded
* Patients with progressive disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria by imaging techniques are not eligible to proceed to the second transplant. Tumor marker increase alone is not sufficient to diagnose disease progression.

Ages: 10 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-12-19 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 Transplants: Patients with Germ Cell Tumors (GCT) treated with a second tandem autologous stem cell transplant (AuSCT) with non-cross-resistant conditioning regimens.
  carboplatin: Days -6, -5, -4: 500mg/m2^/day intravenously (IV) over 60 minutes
  etoposide: 600mg/m^2/day intravenously (IV) over 60 minutes on Days -6 through -3.
  thiotepa: 150mg/m^2/day intravenously IV over 30 minutes; Days -6, -5 and -4
  autologous hematopoietic stem cell transplantation: Peripheral blood stem cell infusion (< 4 x 10^6 CD34+ cells/kg)
  filgrastim: Beginning Day 5, G-CSF 5 μg/kg/day until absolute neutrophil count (ANC) ≥ 1500/UL for 3 consecutive days.
- 1 Transplant: Patients with Germ cell tumors who receive one transplant only.
  ifosfamide: 2500 mg/m^2/day continuous infusion intravenously on Days -6, -5 and -4.
  paclitaxel: 225 mg/m^2 intravenous over 3 hours on Day -7.
  autologous hematopoietic stem cell transplantation: Peripheral blood stem cell infusion (< 4 x 10^6 CD34+ cells/kg)
  Mesna: 2500 mg/m^2/day continuous infusion intravenously on Days -6, -5 and -4.
  filgrastim: Beginning Day 5, G-CSF 5 μg/kg/day until absolute neutrophil count (ANC) ≥ 1500/UL for 3 consecutive days.
Period: Overall Study
Arm/Group | 2 Transplants | 1 Transplant
Started | 14 | 9
Completed | 14 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics collected for the group as a whole prior to decision regarding number of transplants because if a patient did not have enough cells to do two transplants then they only received one transplants.
Groups:
- 2 Transplants/1 Transplant Arms (Overall): Patients with Germ Cell Tumors (GCT) treated with one and second autologous stem cell transplant (AuSCT) with non-cross-resistant conditioning regimens.
Arm/Group | 2 Transplants/1 Transplant Arms (Overall)
Number analyzed (Participants) | 23
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 31 [22 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer. Also called survival rate.
Time Frame: 1 Year
Population: The protocol is essentially one single-arm, but patients received either one or two transplants depending on the cells they had available and we are reporting results for these two groups.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2 Transplants | 1 Transplant
Number analyzed (Participants) | 14 | 9
percentage of participants | 86 [54 to 96] | 56 [20 to 80]

2. Secondary Outcome: Disease-free Survival (DFS)
Description: The number of patients who survive without any signs of symptions of that cancer or any other cancer.
Time Frame: 1 Year
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2 Transplants | 1 Transplant
Number analyzed (Participants) | 14 | 9
percentage of participants | 64 [34 to 83] | 44 [14 to 72]

3. Secondary Outcome: Engraftment of Platelets
Description: Platelet engraftment is defined as 20,000/mm^3 (20 x 10^9/L) for 3 consecutive days unsupported by a platelet transfusion.
Time Frame: Day 100
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 2 Transplants | 1 Transplant
Number analyzed (Participants) | 14 | 9
participants | 13 | 8

4. Secondary Outcome: Numbers of Patients Unable to Mobilize Peripheral Blood Stem Cells
Description: Number of patients unable to achieve adequate stem cell mobilization, need to undergo one or tandem transplantation. Stem cell mobilization = A process in which certain drugs are used to cause the movement of stem cells from the bone marrow into the blood. The stem cells can be collected and stored. They may be used later to replace the bone marrow during a stem cell transplant.
Time Frame: Pre-Transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 2 Transplants | 1 Transplant
Number analyzed (Participants) | 14 | 9
Participants | 0 | 0

5. Secondary Outcome: Engraftment of Neutrophils
Description: Neutrophil engraftment is defined as the first day of three consecutive days where the neutrophil count (absolute neutrophil count) is 500 cells/mm3 (0.5 x 109/L) or greater.
Time Frame: Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 2 Transplants | 1 Transplant
Number analyzed (Participants) | 14 | 9
Participants | 13 | 9

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed for 1 year. Serious and Other (Not Including Serious) Adverse Events monitored/assessed for 100 days after cell infusion.
Description: This trial is single arm study and it is non-randomized. Overall, if patients did not have enough cells to do two transplants then they only received one transplants. This trial is not a two arm protocol.
Groups:
- 2 Transplants/1 Transplant Arms (Overall): Patients with Germ Cell Tumors (GCT) treated with one and second autologous stem cell transplant (AuSCT) with non-cross-resistant conditioning regimens.
  Adverse events are not separable by number of transplants because they were not recorded in to the University of Minnesota's CTMS system. Below you will see AEs for patients with 1 and 2 transplants pooled together.
Arm/Group | 2 Transplants/1 Transplant Arms (Overall)
All-Cause Mortality (participants affected / at risk) | 6/23
Serious Adverse Events (participants affected / at risk) | 8/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Transplants/1 Transplant Arms (Overall) (N=23)
Relapse (Investigations) | 6 (7)
Progressive Disease (Investigations) | 3 (3)
Death (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT00432094/Prot_SAP_000.pdf